CLINICAL TRIAL: NCT02833129
Title: The Effects of Playing High School Football on Later Life Cognitive Functioning and Mental Health: An Observational Study
Brief Title: The Effects of Playing High School Football on Later Life Cognitive Functioning and Mental Health
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Wisconsin, Madison (Other); Moss Rehabilitation Research Institute (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 821703
Record Dates: First submitted 2016-07-07; First posted 2016-07-14 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Memory Impairment; Executive Dysfunction; Depression
MeSH Terms: conditions — Memory Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the effect of playing high school football on later in life cognitive functioning and mental health. This is an observational study that will use data from the Wisconsin Longitudinal Study to compare high school football playing graduates in 1957 with comparable non-high school football playing graduates on cognitive functioning and mental health measures when participants are in their 60s.

DETAILED DESCRIPTION:
The investigators will use data from the Wisconsin Longitudinal Study (WLS) of graduates from Wisconsin high schools in 1957 to investigate the link between playing high-school football and later life depression and cognitive impairment. The WLS has a number of attractive features that make it well-suited for such a study. First, it records whether study participants participated in high school football and also includes detailed measurements of later-life mental health, psychological well-being, and cognition. Second, it includes a rich set of baseline covariates which the investigators will use to construct matched sets of treated and control individuals, including family background, adolescent characteristics, educational and occupational achievement and aspirations. Third, the WLS is one of the few longitudinal data sets that includes an administrative measure of childhood cognition. In short, the WLS provides a large data set that facilitates comparing the later life mental health and cognitive ability of men who played high school football to those who did not, after carefully controlling for a range of potential confounders. The investigators will compare the primary outcomes of the treated subjects to the primary outcomes of the control subjects, after controlling for baseline covariates via full matching with a propensity score caliper. The primary outcomes are depression (modified CES-D score) and cognitive functioning (average of z-scores for letter fluency and delayed word recall) when participants are age 65. Secondary outcomes that include cognitive scores on various domains, the Spielberger anger index, the Spielberger anxiety index and a hostility index will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

-- Male.

Exclusion Criteria:

* No yearbook information available to determine football playing status
* Activity participation in yearbook was not recorded under senior photo or in an index.
* Did not played football but played another high contact sport (soccer, hockey, lacrosse or wrestling).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Graduates of Wisconsin high schools in 1957. The data comes from the Wisconsin Longitudinal Study (WLS), a long-term study of a random sample of 10,317 men and women who graduated from Wisconsin high schools in 1957.
Sampling Method: Probability Sample
Enrollment: 3904 (Actual)
Dates: Start 1957-01; Primary Completion 2003-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Summary score of psychological distress/depression at age 65 | Collected in 2003-2005 when participants were around 65
  Modified CES-D (Center for Epidemiologic Studies Depression Scale) score collected from survey administered when study subjects were approximately 65 years old.
Composite measure of cognition at age 65 | Collected in 2003-2005 when participants were around 65
  Average of the standardized scores from two cognitive functioning tests. In the first test, Letter Fluency, which measures executive functioning, subjects were asked to name as many words beginning with "L" or "F" as they could in 60 seconds. In the second, Delayed Word Recall, which measures memory and attention, subjects were told a list of 10 words and asked to recall as many as possible 12minutes later.

SECONDARY OUTCOMES:
Summary score of psychological distress/depression at ages 54 and 72 | Collected in 1992 and 2011 when participants were around 54 and 72 respectively
  Modified CES-D score collected from surveys administered when study subjects were approximately 54 and 72 years old.
Composite measure of cognition at age 72 | Collected in 2011 when participants were around 72
  Analog of Primary Outcome 2, but based on test results in 2011, when subjects were approximately 72.
Score on Letter Fluency test at ages 65 and 72 | Collected in 2003-2005 and 2011 were around 65 and 72 respectively
  Raw scores on the Letter Fluency test (a component of composite measure of cognition) administered in 2003-05 and 2011.
Score on Delayed Word Recall test at ages 65 and 72 | Collected in 2003-2005 and 2011 when participants were around 65 and 72 respectively
  Raw scores from the Delayed Word Recall test administered in 2003-05 and 2011.
Score on Wechsler Adult Intelligence Scale Similarities test at ages 54, 65, and 72 | Collected in 1992, 2003-2005 and 2011 when participants were around 54, 65 and 72 respectively
  Subjects were asked to describe how two objects from a given list of 9 pairs were alike. Their responses were scored on a fixed scale. For instance, if asked to describe how an orange or a banana are alike, the response "both are fruits" received the highest score (2 points), "both may be eaten" received 1 point, and "both are sweet" received 0 points.
Score on Digit Order test at ages 65 and 72 | Collected in 2003-2005 and 2011 when participants were around 65 and 72 respectively
  Subjects were asked to mentally rearrange and verbally restate increasingly lengthy sets of one-digit numbers such that they are value-ordered from lowest to highest.
Score on McArdle & Woodcock number series test at age 72 | Collected in 2011 when participants were around 72
  Subjects were given a sequence of numbers (e.g. 23, 26, 30, 35, --) and asked to identify the number that correctly completed the sequence. This test is a measure of induction and reasoning, with particular emphasis on quantitative reasoning.
Score on Immediate Word Recall test at ages 65 and 72 | Collected in 2003-2005 and 2011 when participants were around 65 and 72 respectively
  Subjects were read 10 words and asked to immediately recall as many as they can. The same set of words is used in the Delayed Word Recall test.
Hostility index at ages 65 and 72 | Collected in 2003-2005 and 2011 when participants were around 65 and 72 respectively
  Summary measure of subject's hostility based on survey about how he has felt in the week leading up to interview.
Spielberger anxiety index | Collected in 1992, 2003-2005 and 2011 when participants were around 54, 65 and 72 respectively
  Summary measure of subject's anxiety based on survey about how he has felt in the week leading up to interview.
Spielberger anger index | Collected in 1992, 2003-2005 and 2011 when participants were around 54, 65 and 72 respectively
  Summary of subject's anger based on survey about how he has felt in week leading up to interview.
Indicator of heavy drinking status at ages 54, 65, and 72 | Collected in 1992, 2003-05, and 2011 when participants were around 54, 65, and 72, respectively
  A subject is classified as a heavy drinker if he reports having had more than 5 drinks on more than five separate occasions in the month preceding the interview. Based on their responses to the interview, a binary indicator of whether the subject is a heavy drinker was constructed.

OTHER OUTCOMES:
Occupational Prestige Score | Measured in 1975 for jobs held between 1964 and 1975
  Duncan Socioeconomic Index (SEI) scores for the longest job subject held in 1964, 1970, and 1975.
Total earnings | 1974
Indicator of regular, vigorous physical activity at age 35 | Measured in 2011
  Subjects reported whether they regularly engaged in vigorous physical activity at age 35 during the 2011 survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Deshpande, Principal Investigator — University of Pennsylvania; Raiden Hasegawaa, Principal Investigator — University of Pennsylvania; Dylan S Small, PhD, Principal Investigator — University of Pennsylvania

REFERENCES:
- Available data/document: Study Protocol — http://arxiv.org/abs/1607.01756